CLINICAL TRIAL: NCT06074159
Title: Expanding Effective Report-back of Environmental Exposures in Clinic-Based Studies
Brief Title: Impacts of Clinician-Mediated Report-Back
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silent Spring Institute (Other)
Collaborators: University of Puerto Rico (Other); Northeastern University (Other); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1R21ES032934-01A1b; 1R21ES032934-01A1 (NIH)
Record Dates: First submitted 2023-09-14; First posted 2023-10-10 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: All study participants in two pregnancy cohorts will get a personal exposure report for chemicals measured during their pregnancy. 200 participants from each cohort (N Total= 400) are randomly selected and assigned equally to one of two groups: 1) those who only receive their personal results online and 2)those who receive in-clinic to measure differences in participants' environmental health literacy. Pre-and post-tests are administered before and after report-back.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-clinic report-back (Other): 200 participants receive their personal exposure results from a clinician
  Interventions: Behavioral: In-clinic report-back
- Online (Other): 200 participants receive their personal exposure results from a website online
  Interventions: Behavioral: In-clinic report-back

INTERVENTIONS:
Behavioral: In-clinic report-back — Investigators measure whether report-back from a clinician improves environmental health literacy, including leading to greater shifts in exposure-reducing health behaviors

SUMMARY:
The study trains clinicians to return personal exposure results to study participants in pregnancy cohorts, and measures outcomes for environmental health literacy for both clinicians and study participants.

DETAILED DESCRIPTION:
To design and implement clinic-based report-back for endocrine disrupting compounds and analyze the impacts of doing so, investigators train clinicians to report-back individual chemical results to study participants in two pregnancy cohorts and then evaluate outcomes for both clinicians and patients, including shifts in environmental health behaviors, using interviews and pre-and post-tests. All study participants will get a personal exposure report and 200 participants from each cohort (N Total= 400) are randomly selected and assigned equally to one of two groups: 1) those who only receive their personal results online and 2)those who receive them in-clinic to measure additional benefits of clinical report-back for participant learning, exposure-related behaviors, and relationships to the study and clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Participants are of reproductive age

Exclusion Criteria:

* Under 18 years old or past reproductive age

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Environmental health literacy as measured by pre-and post-tests (questionnaires). | 2 weeks
  2 weeks after completing a pre-test and receiving their personal results, study participants will take a post-test. Pre-and post-tests include true and false, as well as scale questions that measure shifts in environmental health literacy before and after report-back.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ohayon, PhD, Principal Investigator — Silent Spring Institute
Locations (2):
- Harvard T.H Chan School of Public Health, Boston, Massachusetts, United States
- University of Puerto Rico Medical Sciences Campus, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No